CLINICAL TRIAL: NCT02309879
Title: Effect of Intravenous Infusion of Lidocaine, Magnesium Sulphate and Remifentanil Perioperatively in Patients Undergoing Mastectomy: a Prospective, Randomized and Double-blind Study
Brief Title: Effect of Infusion of Lidocaine, Magnesium and Remifentanil Perioperatively in Patients Undergoing Mastectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, Fabricio Tavares Mendonca, MD, TSA, Hospital de Base
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LidovsMgvsRemi
Record Dates: First submitted 2014-11-28; First posted 2014-12-05 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Pain
Keywords: Intravenous lidocaine; Magnesium sulphate; Mastectomy; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Remifentanil; Lidocaine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Remifentanil group (Active Comparator): Patients in remifentanil group received an intravenous bolus injection of 2 mg/kg lidocaine followed by a continuous remifentanil infusion of 0,1 mcg/kg/min.
  Interventions: Drug: Remifentanil infusion; Drug: Lidocaine infusion; Drug: Magnesium sulphate infusion; Drug: Magnesium sulphate and Lidocaine infusion
- Lidocaine group (Active Comparator): Patients in lidocaine group received an intravenous bolus injection of 2 mg/kg lidocaine followed by a continuous lidocaine infusion of 3 mg/kg/hr.
  Interventions: Drug: Remifentanil infusion; Drug: Lidocaine infusion; Drug: Magnesium sulphate infusion; Drug: Magnesium sulphate and Lidocaine infusion
- Magnesium group (Active Comparator): Patients in lidocaine group received an intravenous bolus injection of 50 mg/kg magnesium sulphate followed by a continuous magnesium sulphate infusion of 15 mg/kg/hr.
  Interventions: Drug: Remifentanil infusion; Drug: Lidocaine infusion; Drug: Magnesium sulphate infusion; Drug: Magnesium sulphate and Lidocaine infusion
- Magnesium and Lidocaine group (Active Comparator): Patients received an intravenous bolus injection of 2 mg/kg lidocaine plus 50 mg/kg magnesium sulphate followed by a continuous lidocaine infusion of 3 mg/kg/hr plus 15 mg/kg/hr magnesium sulphate
  Interventions: Drug: Remifentanil infusion; Drug: Lidocaine infusion; Drug: Magnesium sulphate infusion; Drug: Magnesium sulphate and Lidocaine infusion

INTERVENTIONS:
Drug: Remifentanil infusion — Patients in Remifentanil group received an intravenous bolus injection of 2 mg/kg lidocaine followed by a continuous remifentanil infusion of 0,1 mcg/kg/min.
  Other Names: Remifentanil hydrochloride
Drug: Lidocaine infusion — Patients in Lidocaine group received an intravenous bolus injection of 2 mg/kg lidocaine followed by a continuous lidocaine infusion of 3 mg/kg/hr.
  Other Names: Lidocaine hydrochloride
Drug: Magnesium sulphate infusion — Patients in Magnesium group received an intravenous bolus injection of 50 mg/kg magnesium sulphate plus an intravenous bolus injection of 2 mg/kg lidocaine followed by a continuous magnesium sulphate infusion of 15 mg/kg/hr.
  Other Names: Magnesium sulphate
Drug: Magnesium sulphate and Lidocaine infusion — Patients in Magnesium and Lidocaine group received an intravenous bolus injection of 2 mg/kg lidocaine plus 50 mg/kg magnesium sulphate followed by a continuous lidocaine infusion of 3 mg/kg/hr plus 15 mg/kg/hr magnesium sulphate
  Other Names: Magnesium sulphate, Lidocaine hydrochloride

SUMMARY:
This study aims to compare the quality of perioperative analgesia of lidocaine, magnesium sulphate and remifentanil in patients undergoing mastectomy

DETAILED DESCRIPTION:
The opioid analgesics are commonly used in clinical practice for pain management in the perioperative period. However, many side effects are associated with its use, such as respiratory depression, nausea, vomiting, drowsiness, itching, urinary retention, constipation, hyperalgesia and impaired immune function. Therefore, alternative techniques and drugs have been used to replace their use. One is the intravenous infusion of lidocaine, a local anesthetic widely used in anesthetic practice. Another is intravenous infusion of magnesium sulphate, a bivalent salt used as a central nervous system depressor, reducing intracranial hypertension, in the treatment of epilepsy; eclampsia; in chronic alcoholism; in hyaline membranes, such as hyperosmotic diuretic; in malnutrition; hypomagnesaemia; in thrombotic microangiopathy; in sickle cell anemia, uterine tetany and atypical ventricular tachycardia. Studies show that the use alone or combined of lidocaine and magnesium sulphate during surgery significantly decreased postoperative pain. The mechanisms of analgesia this local anesthetic in surgical trauma may be blocking neuronal transmission in the lesion site alleviating neurogenic response, and anti-inflammatory systemic intrinsic activity. Intraoperative lidocaine promotes, besides analgesia, decreased consumption of both inhalational anesthetic and opioids; faster return of bowel movements; decreasing the production of interleukins and reduction of airway reactivity. This anesthetic also has significant anti-inflammatory properties, reduces cytokine release both in vitro and in vivo by inhibiting neutrophil activation. N-methyl-D-aspartate (NMDA) receptors are critically involved in the induction and maintenance of neuronal hyperexcitability after traumatic events, therefore, the use of NMDA antagonists before the incision reduces the excitability of the central nervous system and its result is the reduction of clinical hyperalgesia. Magnesium sulphate is an antagonist of glutamate NMDA receptor, which gives analgesic, anticonvulsant and sedative. It acts as a natural physiological calcium antagonist regulating access to the intracellular space. Shows the effect of muscle relaxation by inhibiting the release of acetylcholine at the neuromuscular junction, thereby hypermagnesaemia decreases sensitivity to acetylcholine of the endplate and the potential amplitude endplate. Besides there are few studies with use of these adjuvants during the perioperative period, the intravenous injection of local anesthetic still arouses oddity among professionals; therefore, the investigators interest in the subject.

The patients underwent a prospective, randomized, double blind study, in which the examiners responsible for intra and post-operative will not know which group they were randomly allocated: Lidocaine group (n = 30); Lidocaine and Magnesium group (n = 30); Magnesium group (n = 30) or Remifentanil group (n = 30). Rapid infusion of 0.9% saline 500 ml, in the M and LM group, is added to this solution the loading dose of magnesium sulfate with 50 mg/kg and in group L will only be infused saline 0.9% . Two infusion pumps containing the result of randomization: Lidocaine 3 mg/kg/h and 0.9% saline (L group); magnesium sulphate 15 mg/kg/h and 0.9% saline (M group); lidocaine 3 mg/kg/h and magnesium sulphate 15 mg/kg/hr (LM group); and Remifentanil group (R group).

In the clinical record, the following information will be emphasized: Blood pressure and heart rate intraoperative, perioperative side effects, quantify pain by Visual Analogue Scale (VAS) (ranging from 0 to 10 cm, zero being found when the patient is no pain and ten, with maximum or unbearable pain), Verbal Rating Scale (VRS), consisting of a list of phrases (no pain, mild pain, moderate pain, intense pain, maximum pain) and qualification of pain assessed by the amount of analgesics required postoperatively and the time to request them.

The results were analyzed statistically with the Statistical Package for Social Sciences (SPSS) version 22 (SPSS Inc., Chicago, IL, EUA) using parametric and nonparametric tests, depending on the nature of the variables studied. Data were tested for normality using the Shapiro-Wilk test. Measures of central tendency (means) and dispersion (standard deviation) were used. The level of significance was set at < 0.05. The following tests were used: Mann-Whitney test for age, duration of anesthesia and surgery, time to first analgesic supplementation, total amount of analgesics, pain intensity; Student t-test for weight and height.

ELIGIBILITY:
Inclusion Criteria:

* Female patients scheduled for elective surgery performed mastectomy;
* Physical Status P1 and P2 of the American Society of Anesthesiology (ASA);

Exclusion Criteria:

* Patients with less than 18 years and above 75 years of age;
* Patients who are allergic to morphine and / or lidocaine and / or remifentanil and / or magnesium sulphate;
* Patients with chronic pain;
* Patients with severe hepatic disease;
* Patients with severe renal disease;
* Patients with neurological disorders;
* Patients included in other clinical currently or within the past three months under general anesthesia studies;
* Patients who refuse to participate in the study;
* Any other condition that in the opinion of the investigator, may pose a risk to the patient or interfere with the study objectives;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Analgesics consumption in post-operative | Within the first 24 hours after surgery
  Qualification of pain assessed by the amount of analgesics required postoperatively and the time to request them

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale | Within the first 24 hours after surgery
  Quantify pain by Visual Analogue Scale (VAS, ranging from 0 to 10 cm, zero being found when the patient is no pain and ten, with maximum or unbearable pain)
Pain Scores on the Verbal Rating Scale | Within the first 24 hours after surgery
  Verbal Rating Scale (VRS), consisting of a list of phrases (no pain, mild pain, moderate pain, intense pain, maximum pain)
Anesthetic consumption during surgery | During the surgery
  amount of intravenous and inhalational anesthetics consumed during surgery
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | During the surgery
  Intraoperative hemodynamic stability analysis through the incidence of tachycardia, hypertension, bradycardia, hypotension and consumed vasopressors
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Within the first 24 hours after surgery
  Incidence of adverse effects such as time of awakening, nausea, vomiting, pruritus, urinary retention, drowsiness

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio T Mendonca, MD, TSA, Principal Investigator — Hospital de Base do Distrito Federal, Brazil
Locations (1):
- Hospital de Base do Distrito Federal, Brasília, Federal District, Brazil

REFERENCES:
- [Background] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Derived] Mendonca FT, Pellizzaro D, Grossi BJ, Calvano LA, de Carvalho LSF, Sposito AC. Synergistic effect of the association between lidocaine and magnesium sulfate on peri-operative pain after mastectomy: A randomised, double-blind trial. Eur J Anaesthesiol. 2020 Mar;37(3):224-234. doi: 10.1097/EJA.0000000000001153. PMID 31977625